CLINICAL TRIAL: NCT00238914
Title: Opiate Dependence: Combined Naltrexone/Behavior Therapy
Brief Title: Opiate Dependence: Combined Naltrexone/Behavior Therapy - 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #4260R; R01DA010746 (NIH); R01-10746-1
Expanded Access: Available
Record Dates: First submitted 2005-10-13; First posted 2005-10-14 (Estimated); Last update posted 2012-01-13 (Estimated); Status verified 2012-01

CONDITIONS: Heroin Dependence
MeSH Terms: conditions — Heroin Dependence | interventions — Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CE plus oral naltrexone (Active Comparator): Compliance enhancement plus oral naltrexone
  Interventions: Drug: Naltrexone; Behavioral: Compliance Enhancement (CE)
- BNT plus oral naltrexone (Active Comparator): Behavioral naltrexone therapy plus oral naltrexone
  Interventions: Drug: Naltrexone; Behavioral: Behavioral Naltrexone Therapy (BNT)

INTERVENTIONS:
Drug: Naltrexone — 50mg of oral naltrexone daily
Behavioral: Behavioral Naltrexone Therapy (BNT) — a hybrid of Relapse Prevention, the Community Reinforcement Approach, and Network Therapy
  Arms: BNT plus oral naltrexone
Behavioral: Compliance Enhancement (CE) — a controlled therapy intended to simulate outpatient psychiatric care.
  Arms: CE plus oral naltrexone

SUMMARY:
The overall goal of this research project is to test a newly developed behavioral therapy to enhance the efficacy of naltrexone maintenance and make it a viable alternative to methadone maintenance or detoxification methods for treatment of opiate dependence. HYPOTHESES:

1. Outpatient treatment with Behavioral Naltrexone Therapy will yield a lower rate of relapse to illicit opiates compared to naltrexone plus Compliance Enhancement (CE) Therapy.
2. Lifetime history of depression will predict dysphoria and non-compliance with naltrexone.

DETAILED DESCRIPTION:
Long-term maintenance on naltrexone has proven efficacy as a treatment for opiate dependence, but has not been successful clinically because of at least three problems: 1) The transition from opiate to naltrexone precipitates opiate withdrawal unless the patient has been off any opiates for at least seven days; 2) Compliance issues: patients can miss a few naltrexone doses and begin to experience effects from illicit opiates and become re-addicted, at which point naltrexone cannot be restarted without precipitating withdrawal; 3) Naltrexone may produce dysphoria in some patients. The proposed research study will offer opiate dependent patients brief hospitalization for a rapid detoxification from opiate to naltrexone, using buprenorphine, clonidine and clonazepam. If the patient has already undergone detoxification at an outside unit, they will be assessed for opiate dependence using the naloxone challenge. Patients will then be either discharged or entered directly into outpatient treatment where they will be randomly assigned to either the newly developed "Behavioral Naltrexone Therapy" (BNT), a hybrid of Relapse Prevention, the Community Reinforcement Approach, and Network Therapy or to Compliance Enhancement (CE) therapy, a controlled therapy intended to simulate outpatient psychiatric care. BNT employs behavioral incentives and enlists members of the family and social network to reinforce naltrexone compliance and abstinence. In this current investigation, for both BNT and CE, all patients are maintained on oral naltrexone. Patients are stratified at baseline by presence or absence of lifetime depressive disorder, which the investigators hypothesize will predict dysphoria on naltrexone and non-compliance. Patients are discharged from the hospital, or entered directly, into outpatient treatment at STARS at NYSPI to receive both counseling and Naltrexone, 50 mg per day.

ELIGIBILITY:
Inclusion:

1. Adult, aged 18-60.
2. Meets DSM-IV criteria for current opiate dependence disorder of at least six months duration, supported by a positive urine for opiates and further by a positive naloxone challenge test if the diagnosis is unclear.
3. Able to give informed consent.
4. At least one significant other is willing to be interviewed for possible participation in the treatment.

Exclusion:

1. Pregnancy, lactation, or failure in a sexually active woman to use adequate contraceptive methods.
2. Active medical illness which might make participation hazardous, such as untreated hypertension, unstable cardiovascular disease, acute hepatitis with SGOT or SGPT > 2-3 times normal, unstable diabetes, AIDS dementia.
3. Active psychiatric disorder which might interfere with participation or make participation hazardous, including DSM-IV schizophrenia, bipolar disorder with mania or psychosis, and depressive disorder with suicide risk of 1 or more suicide attempts within the past year.
4. History of allergic reaction to naloxone, naltrexone, buprenorphine, clonidine, or clonazepam.
5. Currently prescribed or regularly taking opiates for chronic pain or medical illness.
6. Current participation in another intensive treatment program or currently prescribed psychotropic medications in the last 30 days.
7. Current participation in a Methadone Maintenance program and/or regular and/or Dependent use of street methadone.
8. Opiate-dependent individuals who are seeking methadone maintenance treatment.
9. History of accidental drug overdose in the last three years as defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 1999-08; Primary Completion 2002-07 (Actual); Study Completion 2002-07 (Actual)

PRIMARY OUTCOMES:
Relapse to heroin addiction | Up to 24 weeks or length of study participation

CONTACTS AND LOCATIONS:
Overall Officials: Edward Nunes, M.D., Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

REFERENCES:
- See also: Related Info — http://www.stars.columbia.edu